CLINICAL TRIAL: NCT03736538
Title: Adjunctive Nitrous Oxide for Acute Suicidal Ideation in Unipolar Depressed Hospitalized Patients
Brief Title: Nitrous Oxide- Suicidal Ideation
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201710183
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder; Depression; Mood Disorders; Suicidal Ideation
Keywords: Nitrous Oxide; Anesthetics
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mood Disorders; Suicidal Ideation | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitrous Oxide (Experimental): Nitrous oxide, an odorless, colorless gas typically used as an induction agent for general anesthesia or for dental sedation, is a known N-methyl-D-aspartate (NMDA) antagonist. It will be given at 50% nitrous oxide/50% oxygen in this study.
  Participants will undergo a maximum of four one hour inhalation sessions as inpatients and 2 booster sessions as outpatients during which they will receive inhaled nitrous oxide.
  Interventions: Drug: Nitrous Oxide
- Placebo Gas (Placebo Comparator): Placebo gas given at 50% nitrogen [inert]/50% oxygen.
  Participants will undergo a maximum of four one hour inhalation sessions as inpatients and 2 booster sessions as outpatients during which they will receive placebo gas.
  Interventions: Drug: Placebo gas

INTERVENTIONS:
Drug: Nitrous Oxide — Nitrous oxide, an odorless, colorless gas typically used as an induction agent for general anesthesia or for dental sedation, is a known N-methyl-D-aspartate (NMDA) antagonist. It will be given at 50% nitrous oxide/50% oxygen in this study.
  Other Names: Laughing Gas
  Arms: Nitrous Oxide
Drug: Placebo gas — Placebo gas given at 50% nitrogen [inert]/50% oxygen.
  Arms: Placebo Gas

SUMMARY:
Most clinical major depression responds to standard treatments (medication and psychotherapy); however, a significant subset of depressed patients (15-20%) do not respond to these treatments and are referred to as treatment-resistant major depression (TRMD). New treatments for TRMD are needed, and one promising line of research are drugs known as N-methyl-D-aspartate (NMDA) glutamate receptor antagonists. In a recent pilot study, the investigators of this study demonstrated that the NMDA antagonist nitrous oxide is effective in TRMD, reducing depressive symptoms, guilt, and suicidal thinking.

To more closely investigate suicidal thinking, this study is designed as a double-blind, randomized, prospective, inpatient trial comparing inhaled nitrous oxide (N2O) plus treatment as usual versus inhaled placebo plus treatment as usual. All unipolar depressed, acutely suicidal inpatients will receive standard treatment for their depression/ suicidal thinking (TAU). Additionally, participants will undergo a maximum of four one hour inhalation sessions as inpatients and 2 booster sessions as outpatients during which they will receive either inhaled nitrous oxide (50% nitrous oxide/50% oxygen = active treatment) or placebo gas (50% nitrogen/50% oxygen). A target total of 50 patients with suicidal ideation and unipolar depression will be enrolled, 25 of whom will be assigned to the TAU control group and 25 of whom will be assigned to the N2O + TAU experimental group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65 years old;
2. current diagnosis of unipolar, major depressive disorder (MDD) without psychosis as defined by the Mini-International Neuropsychiatric Interview (MINI) and The Fourth Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) DSM-IV determined by clinical interview and by a baseline score of ≥18 on the HDRS-21 (Hamilton Depression Rating Scale 21-item;
3. moderate to severe SI defined as a score ≥3 on the HDRS-21 suicide item (item #3);
4. will have good command of the English language;
5. will have been voluntarily admitted to the inpatient Psychiatric Units at Barnes-Jewish Hospital/Washington University in St. Louis, MO.

Exclusion Criteria:

1. Lifetime DSM-IV (obtained via MINI) diagnoses of schizophrenia, schizoaffective disorders, bipolar disorder, obsessive-compulsive disorder, evidence of severe personality disorder (e.g., history of recurrent self-mutilation/cutting, significant and recurrent tumultuous relationships), and panic disorders;
2. past 12-month substance abuse/dependence other than nicotine;
3. active psychotic symptoms;
4. significant pulmonary disease and/or requiring supplemental oxygen;
5. administration of other N-Methyl-D-aspartate (NMDA)-receptor antagonist treatment (e.g., ketamine) within two weeks of entry into study;
6. currently receiving electroconvulsive therapy;
7. contraindications for nitrous oxide (pneumothorax, bowel obstruction, middle ear occlusion, elevated intracranial pressure, chronic cobalamin and/or folate deficiency treated with folic acid or vitamin B12);
8. past 12-month history of head trauma;
9. women who are pregnant or breastfeeding;
10. any other factor that in the investigators' judgment may affect patient safety or compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Severity and number of adverse events in both nitrous oxide and placebo groups | Throughout study duration (approximately 60 days)
  Safety and tolerability of inhaled nitrous oxide will be measured by collecting adverse events in both groups at each study visit throughout the study.
Differential change in suicidal ideation | Baseline to Day 7, approximately 7 days (following the inpatient period inhalation sessions)
  Participants receiving inpatient treatment as usual plus nitrous oxide compared to participants receiving inpatient treatment as usual plus placebo as measured by scores on the 19-item Scale for Suicidal Ideation (SSI; total score range is 0 to 38, higher scores indicate greater suicidal ideation).
Identification of pre-treatment key clinical correlates of anti-suicidal response to nitrous oxide | Change of scores on the SSI for the approximate 7 days of inpatient period
  Correlations of change in Scale for Suicidal Ideation score (SSI; total score range is 0 to 38, higher scores indicate greater suicidal ideation) at end of inpatient period with: 1) presence of family history of alcohol dependence; 2) a personal/family history of suicide attempt or a family history of suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Conway, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States